CLINICAL TRIAL: NCT02133170
Title: Comparative Efficacy of Two Adjunctive Psychosocial Interventions (Mindfulness or Psychoeducation) Versus Treatment as Usual in Bipolar Patients With Subsyndromal Deppresive Symptoms: A Pilot Randomized Trial
Brief Title: "Mindfulness vs Psychoeducation in Bipolar Disorder"
Acronym: BI-MIND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HULP: 4094
Record Dates: First submitted 2014-04-30; First posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Bipolar; Depressive Symptoms
Keywords: BIPOLAR DISORDER; DEPRESSIVE SYMPTOMS; MINDFULNESS; PSYCHOEDUCATION; BIPOLAR PATIENTS WITH DEPRESSIVE SYMPTOMS
MeSH Terms: conditions — Depression; Bipolar Disorder | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Psychopharmacological + MBCT (Active Comparator): psychopharmacological treatment plus Mindfulness Based Cognitive Therapy (MBCT)
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy (MBCT)
- psychopharmacological + psychoeducation (Active Comparator): psychopharmacological treatment plus structured group psychoeducation;
  Interventions: Behavioral: Psychoeducation
- Psychopharmacological treatment. (Other): Treatment as usual (TAU), including standard psychiatric care with psychopharmacological treatment.
  Interventions: Behavioral: Standard treatment

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy (MBCT) — The MBCT program is conducted in HULP (BRV and CBP), which also train therapists from Vitoria, in order to homogenize the intervention. Random sessions are video or audio recorded to be discussed and analyzed by the treatment team. The manualized MBCT therapy consists of 8 weekly sessions of 90 minutes and is applied in groups of approximately 10-15 patients. At least two programs in H. La Paz and two in the hospital de Santiago (Vitoria) will be provided.
  Arms: Psychopharmacological + MBCT
Behavioral: Psychoeducation — Psychoeducation program will be held in groups of 10 to 15 patients in 90-minute weekly sessions led by two therapists also outside the research team. The specific program of 8 sessions is focused addressing disease awareness, adherence to treatment and early detection of prodromal symptoms. Homework will also be included. The program is based on the Psychoeducation Manual for Bipolar Disorder . F.Colom , E.Vieta . Ars Medica, 2004. Attendance at least 80 % of the sessions of both interventions will be required to be considered complete.
  Arms: psychopharmacological + psychoeducation
Behavioral: Standard treatment — Treatment as usual (TAU), including standard psychiatric care with psychopharmacological treatment.
  Arms: Psychopharmacological treatment.

SUMMARY:
This is a parallel 3-group, multicenter, prospective, randomized, single-blind (evaluator) controlled pilot trial, with a 38- week follow-up. Patients diagnosed with bipolar disorder (BD) according to DSM -5 criteria for mild depression or subsyndromal depressive symptoms are assigned to one of the following 3 treatment groups: 1) psychopharmacological treatment plus Mindfulness Based Cognitive Therapy (MBCT); 2) psychopharmacological treatment plus structured group psychoeducation; 3) treatment as usual (TAU), including standard psychiatric care with standard pharmacologic treatment.

DETAILED DESCRIPTION:
This is a parallel 3-group, multicenter, prospective, randomized, single-blind (evaluator) controlled pilot trial, with a 38- week follow-up. Patients diagnosed with bipolar disorder (BD) according to DSM -5 criteria for mild depression or subsyndromal depressive symptoms are assigned to one of the following 3 treatment groups: 1) psychopharmacological treatment plus Mindfulness Based Cognitive Therapy (MBCT); 2) psychopharmacological treatment plus structured group psychoeducation; 3) treatment as usual (TAU), including standard psychiatric care with standard pharmacologic treatment. After written informed consent is signed, patients meeting the inclusion criteria are randomized (2:2:1 ratio) through a Random Allocation Software. All three groups are assessed at baseline (t0), immediately after completing the program (t1; 8 weeks) and at follow-up six months after randomization. The assessments include the following variables: depression, anxiety, general and social cognition, global functioning, BDNF, and other clinical variables. The evaluator who collected the biomarkers and the clinical and psychometric data will be blind to treatment. The interrater variability between all researchers will be checked.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years
* BD type I or II, in clinical remission of acute mood episode at least in the three months prior to study
* Having presented an acute affective episode in the past 3 years
* Having presented at least two depressive episodes throughout his life.
* Monotherapy or combination with a mood stabilizer (lithium, valproate, carbamazepine or lamotrigine) at optimal doses (ie, in serum levels within the therapeutic range: 0.6-1.2 mEq / L for lithium, 50-100 ug / ml for valproate, and 5-12 mcg / mL for carbamazepine), or quetiapine monotherapy or in combination with the aforementioned stabilizers, or any oral atypical antipsychotic in combination with an antidepressant
* Hamilton Depression Rating Scale [HDRS]-17 score ≥ 8 and ≤ 19 and Young Mania Rating Scale [YMRS] score <8
* Being able to understand and comply with the requirements of the trial
* Written consent to participate in the study.

Exclusion Criteria:

* Any acute mood episode in the 12 weeks before the start of the trial.
* Any current DSM -5 diagnosis different from bipolar disorder (including substance or alcohol use disorder at the time of study entry, except if it is under complete remission. Not applicable to nicotine or caffeine)
* Risk of suicide or self/hetero aggressiveness
* Pregnancy
* Severe and unstable medical pathology.
* Patients who are currently receiving structured psychotherapy or structured group psychoeducation about bipolar disorder, or who have received structured psychoeducation in the past 5 years
* Patients who are treated with a different mood stabilizer to lithium , valproate , carbamazepine , lamotrigine, a classic antipsychotic or antidepressant monotherapy at the time of the randomization
* Treatment with a depot antipsychotic
* Participation in another clinical trial within 4 weeks prior to randomization
* Mental Retardation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint of the study is given by changes in the overall score of the Hamilton Rating Scale for Depression (HDRS) | from baseline (V0) to week 8 (V1)
  Primary endpoint of the study is given by changes in the overall score of the Hamilton Rating Scale for Depression (HDRS), from baseline (V0) to week 8 (v1) for each of the treatment groups.

SECONDARY OUTCOMES:
Changes in the global score of Young Mania Rating Scale (YMRS) | from baseline (V0) to week 8 (V1)
  Changes in the global score of Young Mania Rating Scale (YMRS) from baseline (V0) to visit 1 (at the end of surgery 8 weeks (v1)
Changes in scale score of Clinical Global Impression CGI-BP | from baseline (V0) to week 8 (V1)
  Changes in scale score of Clinical Global Impression CGI-BP from baseline (V0) to visit 1
Changes in the score of the Hamilton Rating Scale for Anxiety HAM-A | from baseline (V0) to week 8 (V1)
  Changes in the score of the Hamilton Rating Scale for Anxiety HAM-A from baseline (V0) to visit 1
Cognitive changes | from baseline (V0) to week 8 (V1)
  Changes at the end of the intervention will be assessed with the following measures:
  * sustained and selective attention
  * working memory and executive functions
  * perception of the attitude of mindfulness ( FFMQ ) in patients in the experimental group
  * scales of social cognition
Functioning | from baseline (V0) to week 8 (V1)
  Changes in total scale score of the Functioning Assessment Short Test (FAST)
Plasmatic levels of Brain-Derived Neurotrophic Factor (BDNF): | from baseline (V0) to week 8 (V1)
  Plasmatic levels of Brain-Derived Neurotrophic Factor (BDNF): changes from baseline to visit 1
Recurrence | from baseline (V0) to week 8 (V1)
  Recurrence, defined as the emergence of a new acute episode whether depressive, mixed, hypo or manic at any time throughout the study, according to DSM-5 clinical criteria or when the score on the HDRS scale is ≥ 20 ( depressive episode ) or the Young scale ( YMRS ≥ 8) (hypo/manic episode), or a change drug or hospitalization is needed.

OTHER OUTCOMES:
changes in the overall score of the Hamilton Depression Rating Scale (HDRS ) | from baseline (V0 ) to week 24 (V2)
  Changes in the overall score of the Hamilton Depression Rating Scale (HDRS ) from baseline (V0 ) to week 24 (V2)
Changes in the Young Mania Rating Scale (YMRS) | from baseline (V0 ) to week 24 (V2)
  Changes in the Young Mania Rating Scale (YMRS) from baseline (V0 ) to week 24 (V2)
Changes in the overall score of the Hamilton anxiety Scale HAM- A | from baseline (V0 ) to week 24 (V2)
  changes in the overall score of the Hamilton anxiety Scale HAM- A from baseline (V0 ) to week 24 (V2)
Cognitive changes | from baseline (V0 ) to week 24 (V2)
  Cognitive changes: changes at the end of the intervention will be assessed with the following measures:
  * sustained and selective attention
  * working memory and executive functions
  * perception of the attitude of mindfulness ( FFMQ ) in patients in the experimental group
  * scales of social cognition
Functioning: | from baseline (V0 ) to week 24 (V2)
  Functioning: changes in total scale score of the Functioning Assessment Short Test (FAST)
Plasmatic levels of Brain-Derived Neurotrophic Factor (BDNF) | from baseline (V0 ) to week 24 (V2)
  Plasmatic levels of Brain-Derived Neurotrophic Factor (BDNF): changes from baseline to visit 2
Plasmatic levels of Brain-Derived Neurotrophic Factor (BDNF): | from baseline (V0) to week 8 (V1)
  Plasmatic levels of Brain-Derived Neurotrophic Factor (BDNF): changes from baseline to visit 1 (end of intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Consuelo De Dios Perrino, MD PhD, Principal Investigator — Hospital Universitario La Paz
Locations (2):
- Spain (2):
  - Hospital Santiago Apostol, Vitoria-Gasteiz, Alava
  - Hospital Universitario La Paz, Madrid, Madrid

REFERENCES:
- [Derived] Carracedo-Sanchidrian D, de Dios-Perrino C, Bayon-Perez C, Rodriguez-Vega B, Bravo-Ortiz MF, Ortega MA, Gonzalez-Pinto AM, Lahera G. Effect of mindfulness-based cognitive therapy vs. psychoeducational intervention on plasma brain-derived neurotrophic factor and cognitive function in bipolar patients: a randomized controlled trial. Front Psychiatry. 2024 Jan 5;14:1279342. doi: 10.3389/fpsyt.2023.1279342. eCollection 2023. PMID 38250270
- [Derived] Lahera G, Bayon C, Fe Bravo-Ortiz M, Rodriguez-Vega B, Barbeito S, Saenz M, Avedillo C, Villanueva R, Ugarte A, Gonzalez-Pinto A, de Dios C. Mindfulness-based cognitive therapy versus psychoeducational intervention in bipolar outpatients with sub-threshold depressive symptoms: a randomized controlled trial. BMC Psychiatry. 2014 Aug 15;14:215. doi: 10.1186/s12888-014-0215-x. PMID 25124510
- See also: Related Info — http://idipaz.es